CLINICAL TRIAL: NCT02140840
Title: A Phase II Open-Label, Multiple-Dose, Single Agent Study to Evaluate the Overall Response Rate of Orally Administered Trametinib in Patients With Relapsed of Refractory Multiple Myeloma
Brief Title: UARK 2014-08 A Phase II Open-Label, Multiple-Dose, Single Agent Study to Evaluate the Overall Response Rate of Orally Administered Trametinib
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202550
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Myeloma
Keywords: TMTB; Mekinist; Trametinib; relapse; refractory; response rate
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Trametinib — 2 mg of Trametinib daily by mouth in 28 day cycles
  Other Names: Mekinist; TMTB; JTP-74057; JTP-78296; JTP-75303

SUMMARY:
The purpose of this study is to evaluate the overall response rate of Trametinib when administered orally to patients with relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
The effect of on tumor response will be determined using the International Myeloma Working Group uniform response criteria by analyzing changes in serum and urine values of monoclonal protein immunoglobulin kappa and lambda free light chain and ratio, microglobulin, lactate dehydrogenase, hemoglobin and C-reactive proten.

ELIGIBILITY:
Inclusion Criteria:

* Been identified as having multiple myeloma with activating NRAS, KRAS or BRAF genetic mutations on CD138+ cells, identified by molecular genetic testing
* Have been diagnosed with multiple myeloma by having met all three of the following IMWG criteria:

a Clonal bone marrow plasma cells >10% b Presence of serum and/or urinary M-protein (If no monoclonal protein is detected (non-secretory disease), then >/= 30% monoclonal bone marrow plasma cells and/or a biopsy-proven plasmacytoma required.) c Evidence of end-organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically, one or more of the following: (i) Hypercalcemia: serum calcium >11.5 mg/100 mL (ii) Renal insufficiency: serum creatinine >2 mg/dL (iii) Anemia: normochromic, normocytic with a hemoglobin value >2 g/100 mL below the lower limit of normal or a hemoglobin value <10 g/100 mL (iv)Bone lesions: lytic lesions, severe osteopenia, or pathologic fracture.

* Have measurable disease defined by the following:

  (i) Serum M-protein ≥1g/dL or urine M-protein ≥200 mg/24 hours by protein electrophoresis (ii) If neither serum nor urine M-protein meet the criteria above, then kappa or lambda serum FLC must be ≥10 mg/dL accompanied by an abnormal kappa to lambda ratio (<0.26 or >1.65) (Serum FLC should only be used for patients without measurable serum or urine M-protein spike.)
* Have relapsed or refractory disease after two or more prior multiple myeloma treatment regimens, each of which may have consisted of either single or multiple therapies
* Be at least 3 weeks beyond the last multiple myeloma therapy and have recovered from acute toxicities of prior therapies measured by CTCAE Ver 3.0.
* Have an Eastern Cooperative Oncology Group performance status of 0 to 2
* Have life expectancy of at least 3 months
* Be ≥18 years of age and willing to provide written informed consent
* For women of childbearing potential, must have used effective contraceptive methods for previous 4 weeks and agree to continue using such methods during the study and for at least 4 months after completing the study, this must include the use of a male/female latex barrier method of contraception (for male participants (See APPENDIX K). TMTB is a pregnancy category D drug. A female of childbearing potential is defined as a female who has not been in natural menopause for the previous, consecutive 24 months, or undergone hysterectomy or bilateral oophortectomy. Women of childbearing potential must have a negative serum pregnancy test within 24 hours before the initiation of TMTB therapy.
* Have an absolute neutrophil count >1,000/mm3
* Have a platelet count >50,000/mm3
* Have total direct bilirubin <2.0 mg/dL
* Have aspartate aminotransferase and alanine aminotransferase ≤3 times the upper limit of normal
* Have serum creatinine ≤2.5 times the upper limit of normal
* Have hemoglobin ≥8.5 g/dL
* All prior treatment- related toxicities must be CTCAE (Version 3.0) ≤ Grade 1 (except alopecia)
* Subject is able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels

Exclusion Criteria:

* Have an active infection or serious comorbid medical condition
* Be receiving other concurrent anticancer agents or therapies
* Be receiving other concurrent investigational therapies or have received investigational therapies within 3 weeks of screening, not inclusive of molecular genetic testing
* Be eligible to receive any other standard therapy available that is known to extend life expectancy
* For women be pregnant, nursing, unwilling or unable to utilize two forms of birth control, including the use of a latex condom.
* Have a history of another malignancy, except as noted below Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer and/or subjects with indolent second malignancies are eligible.
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* History of interstitial lung disease or pneumonitis.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to randomization and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to randomization.
* History of retinal vein occlusion (RVO)
* Symptomatic or untreated spinal cord compression.
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted).
* History or evidence of cardiovascular risk including any of the following (See APPENDIX M for more details):

a LVEF<LLN b A QT interval of ≥ 480 msec corrected for heart rate using the Bazett's formula (QTcB;).

c History or evidence of current clinically significant uncontrolled arrhythmias.

Exception: Subjects with controlled atrial fibrillation for >30 days prior to study enrollment d History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study enrollment

* History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association (NYHA).

a Treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy; b Patients with intra-cardiac defibrillators; c Known cardiac metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The response rate of Trametinib when administered orally to patients with relapsed multiple myeloma | 28 day

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heuck, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States